CLINICAL TRIAL: NCT01065090
Title: A Single-blinded, Controlled, Multi-centre Study of Effects of Exercise in Patients With Multiple Sclerosis
Brief Title: A Single-blinded, Controlled, Multi-centre Study of Effects of Exercise in Participants With Multiple Sclerosis
Acronym: ACTIMS
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Collaborators: Biogen Idec A/S (Unknown)
Responsible Party: Sponsor
Other Study IDs: ACTIMS
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Exercise
Keywords: Capacity for Work Questionnaire; exercise; AVONEX; SDMT: Symbol Digit Modalities Test; FSMC: Fatigue Scale for Motor and Cognitive functions; effects of exercise; EDSS: Expanded Disability Status Scale
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- training: one group will receive resistance training and one group the normal physiotherapeutic treatment
- physiotherapy: one group will receive resistance training and one group the normal physiotherapeutic treatment

SUMMARY:
The primary objective of the investigation is to determine whether the addition of exercise (resistance training or modified physiotherapy) improves functional capacity in Multiple Sclerosis (MS) participants undergoing Disease Modifying Therapy (DMT) treatment. We hypothesize that the Progressive Resistance Training (PRT) will improve functional capacity without increasing the risk of relapses in participants undergoing standard DMT treatment. The secondary objectives are to determine whether exercise (resistance training or physiotherapy) improves fatigue, mood and Quality of Life (QoL) in MS participants undergoing DMT treatment. Also as a secondary objective, the study aims at determining whether exercise (resistance training or modified physiotherapy) has an impact on Expanded Disability Status Scale (EDSS), time to first relapse, number of relapse free participants, and immunological factors. We hypothesize that the exercise (resistance training) will improve fatigue, mood and QoL and that an impact on immunological factors will be seen in participants even though they are undergoing standard DMT treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Age > 18 years and age < 65 years at screening
* Relapsing Remitting Multiple Sclerosis (RRMS) diagnosis according to McDonald Criteria
* Subjects who have been on Avonex treatment for 3-6 months prior to screening
* A signed informed consent form (ICF) is obtained before any study activity
* EDSS > 1.5 and < 5 at Screening with at least a score of 1 in pyramidal function
* Are able to walk at least 100 meters
* Are able to transport themselves to and from the training facility

Key Exclusion Criteria:

* Suffer from dementia, alcoholism or if they use pacemaker
* Have any serious medical co-morbidities like cardiovascular, respiratory, orthopedic or metabolic diseases
* Have had a MS relapse within an eight week period prior to the study start
* Are pregnant
* Have trained systematic resistance training for one day or more each week in the prior 3 months before study start.
* Only able to participate in less than 70% of the planned training sessions.
* Suffers from major depression

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients on AVONEX 3-6 months after treatment initiation
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2010-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change of muscle strength | Baseline, 12 months, 15 months and 18 months.
  Measured by chair stand test

SECONDARY OUTCOMES:
Changes of speed of walking | Baseline, 12 months and 18 months
  Measured by 6 min walk test, Symbol Digit Modalities Test (SDMT), Quality of Life (QoL, SF26, physical part) and Multiple Sclerosis Walking Scale (MSWS)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (14):
- Coordinating Research Site, NSW, Australia
- Denmark (3):
  - Research Site, Odense
  - Research Site, Sønderborg
  - Research Site, Vejle
- Finland (4):
  - Research Site, Jyväskylä
  - Research Site, Oulu
  - Research Site, Pori
  - Research Site, Seinäjokï
- Research Site, Hamilton, New Zealand
- Norway (2):
  - Research Site, Drammen
  - Research Site, Ullevål
- Sweden (3):
  - Research Site, Ängelholm
  - Research Site, Gothenburg
  - Research Site, Stockholm